CLINICAL TRIAL: NCT00803153
Title: Pattern Scan Laser Photocoagulation: Safety and Complications, Experience After 1301 Consecutive Cases.
Brief Title: PASCAL: Safety and Complications, Experience After 1301 Consecutive Cases
Status: Withdrawn | Type: Observational
Why Stopped: undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Other Study IDs: APEC-038
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Bruch Rupture; Choroidal Detachment
Keywords: Panretinal photocoagulation; Bruch rupture; Choroidal detachment; complication rates
MeSH Terms: conditions — Choroidal Effusions | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Panretinal Photocoagulation [Pattern Scan Laser (PASCAL) system]

SUMMARY:
To report the safety and incidence of adverse effects, during and after a successful photocoagulation for different pathologies using a Pattern Scan Laser (PASCAL) system and its modified settings

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with PASCAL system

Exclusion Criteria:

* Uncompleted file.
* Loss of follow-up.

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients which has been treated with the pattern scan laser system between november 2007 to july 2008.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Complication rates | during treatment and follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación para Evitar la Ceguera en México, Mexico City, Mexico City, Mexico